CLINICAL TRIAL: NCT02505477
Title: Mechanisms of Improving Cognition and Negative Symptoms in Schizophrenia With N-Acetylcysteine: a Magnetic Resonance Spectroscopy Study of Glutamate and Glutathione
Brief Title: Treatment of Cognitive and Negative Symptoms in Schizophrenia With N-acetylcysteine
Acronym: NAC2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FOS53929
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Schizophrenia; Cognitive Deficits; Schizophrenia; Negative Type
Keywords: schiozphrenia; cognition; negative symptoms; glutamate; glutathione; N-acetylcysteine
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — Acetylcysteine; Cysteine; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine (Experimental): Patients in this group will receive N-acetylcysteine (NAC) 1200mg orally twice daily (total daily dose 2400mg), for eight weeks. Each individual tablet contains 300mg NAC, therefore patients will take two tablets by mouth each morning and two tablets by mouth each evening. Manufacturer: Jarrow Industries, Inc.; Brand name: N-A-C Sustain
  Interventions: Drug: N-acetylcysteine; Other: Treatment as Usual
- Placebo (Placebo Comparator): Patients in this group will receive placebo tablets indistinguishable from NAC tablets, with the same protocol as NAC: two placebo tablets by mouth each morning, and two placebo tablets by mouth each evening. Manufacturer: Jarrow Industries, Inc.; Brand name: N-A-C Sustain
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine is a safe, widely available supplement currently FDA-approved for treatment of acetaminophen antidote and as a mucolytic. It has effects on glutamate in the brain via the NMDA receptor as well as the glutathione antioxidant system (it is a precursor to glutathione).
  Other Names: NAC, acetylcysteine, cysteine, Acetadote
  Arms: N-acetylcysteine
Other: Treatment as Usual — Treatment for schizophrenia which may include medications, therapy, or other types of treatment as determined by the subject's VA or community psychiatrist or mental health treatment team

SUMMARY:
The purpose of this study is to attempt to treat cognitive and negative symptoms of schizophrenia, with the nutritional supplement N-acetylcysteine (NAC).

Schizophrenia is a chronic mental disorder that affects approximately 65 million people worldwide, and causes significant disability and suffering. Patients with schizophrenia often hear voices and have persecutory delusions. Though these are the most recognizable features of the illness, the deficits most closely linked to disability are known as cognitive deficits and negative symptoms. Cognitive abilities refer to the ability to perform mental tasks that require focus and attention, and also include memory and verbal skills. Negative symptoms refer to a lack of interest in the world, and decreased social interactions. In our study, the investigators aim to improve these symptoms and deficits by targeting the glutamate system.

Glutamate is the major excitatory neurotransmitter in the brain, and its regulation is abnormal in schizophrenia: glutamate levels are too low at some receptors, and too high at others. As well, free radicals surrounding glutamate receptors also interfere with their proper function. N-acetylcystine (NAC) is a safe and widely-available dietary supplement that may restore glutamate to its correct levels in the brain, and may also help protect the brain from antioxidant damage.

In our study, patients with schizophrenia will be randomly assigned to receive either NAC or placebo for 8 weeks. Brain levels of glutamate and an important antioxidant, glutathione, will be measured before and after treatment, using a neuroimaging technique known as magnetic resonance spectroscopy. Cognitive and negative symptoms will also be assessed before, during and after treatment. The investigators hypothesize that glutamate and glutathione will be normalized in patients' brains, and that their negative and cognitive symptoms will be improved, too.

DETAILED DESCRIPTION:
Schizophrenia is a severe mental illness associated with hallucinations and delusions (positive symptoms), emotional withdrawal and decreased expressivity (negative symptoms), and problems with memory, attention, and social interaction (cognitive impairment). Positive symptoms, the most recognizable characteristics of the illness, can be treated effectively with available antipsychotic medications. Cognitive deficits and negative symptoms, however, are more closely related to functional outcome in schizophrenia, and yet, there is no approved treatment for these types of deficits (1,2).

One prominent theory proposes that these deficits and symptoms arise from dysfunctional receptors for the major excitatory neurotransmitter in the brain, glutamate (3), in two different ways. First, it is believed that decreased signaling from glutamate receptors on inhibitory neurons leads to excessive glutamate activity in the prefrontal cortex, resulting in cognitive impairment (2). This decreased signaling from glutamate receptors may result from too little glutamate present at receptors with mGlu2/3 subunits on inhibitory neurons. In a second mechanism, excessive oxidizing species surrounding glutamate receptors in schizophrenia cause receptor hypofunction (2). Glutathione, the most important protective molecule against oxidative stress in the brain, is protective against this. Importantly, glutathione was found to be 52% lower in medial prefrontal cortex of schizophrenia patients compared to controls (4). In rats, inhibition of glutathione synthesis produced cognitive deficits, and a recent study showed an inverse correlation between glutathione and negative symptoms in patients (5,6). Remarkably, there is an agent that affects both glutamate and glutathione: the dietary supplement N-acetylcysteine, or NAC.

NAC is a safe and widely available dietary supplement that may be able to alter the pathophysiology of schizophrenia by affecting both glutamate and glutathione. Within the glutamate system, NAC acts on inhibitory neurons to restore inhibitory tone on glutamatergic neurons in the frontal cortex (7). A study published in 2012 showed NAC normalized glutamate levels in cingulate cortex of cocaine-dependent patients (8). Remarkably, NAC is also the precursor to glutathione, and NAC administration increases serum glutathione concentrations (9,10). In one randomized, placebo-controlled study, NAC administration correlated with improvement in negative symptoms in schizophrenia patients (11). We propose to investigate the mechanisms of the putative therapeutic benefit of NAC for patients with schizophrenia, and to explore its impact on negative symptoms and cognition.

In this study, we will use magnetic resonance spectroscopy (MRS) to measure glutamate levels in prefrontal cortex, hypothesizing that NAC will normalize, and therefore reduce, levels of glutamate. We will measure glutathione levels with both MRS and serum levels, hypothesizing that NAC will increase glutathione levels in the brain and systemically. We will measure negative symptoms before, during and after treatment with NAC, hypothesizing an improvement in the NAC treatment group compared to placebo, based on findings in the literature. Finally, as an exploratory aim, we will measure performance on the MATRICS Consensus Cognitive Battery (MCCB), before and after NAC treatment, to test effects of NAC on cognition in schizophrenia.

In 40 subjects with a diagnosis of schizophrenia or schizoaffective disorder, we will conduct a randomized, double-blind, placebo-controlled study with NAC (total daily dose 2400mg) or placebo over an 8-week period.

* Specific Aim 1: Compare glutamate in bilateral dorsolateral prefrontal cortex before and after NAC vs. placebo treatment using MRS

  o Hypothesis 1: Prefrontal glutamate concentration will be normalized (reduced) after treatment with NAC, but not after treatment with placebo.
* Specific Aim 2: Compare glutathione in medial prefrontal cortex before and after NAC vs. placebo treatment using MRS

  * Hypothesis 2a: Medial prefrontal cortical glutathione concentration will be improved (increased) after treatment with NAC, but not placebo
  * Hypothesis 2b: Serum glutathione levels will be increased after treatment with NAC, but not placebo
* Specific Aim 3: Compare negative symptoms before, during and after NAC vs. placebo treatment

  o Hypothesis 3: Negative symptoms will be improved after treatment with NAC, but not placebo
* Exploratory Aim: Assess performance on the MCCB before and after treatment with NAC vs. placebo

References

1. Green, M. F. & Nuchterlein, K. H. Should Schizophrenia Be Treated as a Neurocognitive Disorder? Schizophrenia bulletin 25, 309-318 (1999).
2. Moghaddam, B. & Javitt, D. From Revolution to Evolution: The Glutamate Hypothesis of Schizophrenia and its Implication for Treatment. Neuropsychopharmacology 37, 4-15 (2011).
3. Moghaddam, B. Targeting metabotropic glutamate receptors for treatment of the cognitive symptoms of schizophrenia. Psychopharmacology (Berl) 174, (2004).
4. Do, K. Q. et al. Schizophrenia: glutathione deficit in cerebrospinal fluid and prefrontal cortex in vivo. European Journal of Neuroscience 12, 3721-3728 (2000).
5. Castagné, V., Rougemont, M., Cuenod, M. & Do, K. Q. Low brain glutathione and ascorbic acid associated with dopamine uptake inhibition during rat's development induce long-term cognitive deficit: relevance to schizophrenia. Neurobiology of Disease 15, 93-105 (2004).
6. Matsuzawa, D. et al. Negative Correlation between Brain Glutathione Level and Negative Symptoms in Schizophrenia: A 3T 1H-MRS Study. PLoS ONE 3, e1944 (2008).
7. Berk, M., Malhi, G. S., Gray, L. J. & Dean, O. M. The promise of N-acetylcysteine in neuropsychiatry. Trends in Pharmacological Sciences 34, 168-178 (2013).

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-5 criteria for schizophrenia or schizoaffective disorder
* Must be able to provide informed consent to participate in the research project

Exclusion Criteria:

* Actively participating in other experimental drug trial(s) either currently or within the past month
* Psychiatric hospitalization within the previous three months
* Medical hospitalization or other acute medical problem within the previous three months
* A greater than 50% change in dose of antipsychotic medication within the previous three months
* They have met DSM-5 criteria for substance use disorder within the previous three months
* History of neurological illness including stroke, epilepsy, or loss of consciousness for 60 minutes or more

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Improvement of negative symptoms | 0 weeks (baseline), 4 weeks and 8 weeks of treatment with NAC
  Negative symptoms will be assessed with the PANSS and the CAINS
Glutamate levels in prefrontal cortex | 0 weeks (baseline) and 8 weeks of treatment with NAC
  Patients will undergo a magnetic resonance spectroscopy scan to measure glutamate levels in prefrontal cortex
Glutathione levels in prefrontal cortex | 0 weeks (baseline) and 8 weeks of treatment with NAC
  Patients will undergo a magnetic resonance spectroscopy scan to measure glutathione levels in prefrontal cortex

SECONDARY OUTCOMES:
Whole blood glutathione level | 0 weeks (baseline) and 8 weeks of treatment with NAC

OTHER OUTCOMES:
Cognitive Performance on the MCCB | 0 weeks (baseline) and 8 weeks of treatment with NAC
  Patients will be evaluated for performance on the Matrics Consensus Cognitive Battery

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Yang, MD, PhD, Principal Investigator — Assistant Clinical Professor
Locations (1):
- UCLA Semel Institute for Neuroscience and Human Behavior, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No